CLINICAL TRIAL: NCT03175198
Title: Post-Marketing Surveillance on the Use of Prazaxa® Capsules in Japanese Patients With Nonvalvular Atrial Fibrillation After the Availability of Idarucizumab
Brief Title: Japanese Pradaxa PMS, Long Term
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160-0284
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Results first posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with nonvalvular atrial fibrillation (NVAF): Patients with nonvalvular atrial fibrillation (NVAF) taking daily oral dose of Prazaxa® Capsules (Dabigatran etexilate). Dosage of Dabigatran etexilate approved in Japan: 300 milligram (mg) daily (150 mg [as 2 capsules of 75 mg] twice a day (b.i.d)) or 220 mg (110 mg [as 1 capsule of 110 mg] b.i.d) for a treatment duration of 52 weeks.
  Interventions: Drug: Prazaxa® Capsules

INTERVENTIONS:
Drug: Prazaxa® Capsules — Dosage of Dabigatran etexilate approved in Japan: 300 milligram (mg) daily (150 mg [as 2 capsules of 75 mg] twice a day (b.i.d)) or 220 mg (110 mg [as 1 capsule of 110 mg] b.i.d) for a treatment duration of 52 weeks.
  Other Names: Dabigatran etexilate

SUMMARY:
The study objective is to confirm appropriate use and safety profile of Prazaxa® Capsules in real-world setting after the availability of idarucizumab

DETAILED DESCRIPTION:
The study is Post-Marketing Surveillance on the Long-Term Use of Prazaxa® Capsules in Japanese patients with nonvalvular atrial fibrillation after the availability of idarucizumab. Even after the availability of idarucizumab in real clinical practice, appropriate use of Prazaxa® Capsules will continue. The patient population who receive Prazaxa® Capsules and the safety profile of Prazaxa® Capsules is not expected to change. This study investigates appropriate use with prospective investigation in the routine medical practice

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with nonvalvular atrial fibrillation who have never received Prazaxa® Capsules / dabigatran etexilate for preventing the occurrence of ischemic stroke and systemic embolism before enrolment in Japan

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An observational study, no specific treatment is mandated or withheld from the patients. The choice of maintenance treatment for nonvalvular atrial fibrillation must be according to regular medical practice and at discretion of physician (i.e., no randomised assignment of patient to treatment [Prazaxa® Capsules or other treatment] is performed).
Sampling Method: Non-Probability Sample
Enrollment: 5660 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rie Ikeda, 81364172200, Study Chair — zzCDMJP_PV_PMS@boehringer-ingelheim.com
Locations (1):
- Nippon Boehringer Ingelheim Co., Ltd, Tokyo, Japan

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Post-Marketing Surveillance on the Long-Term Use of Prazaxa® Capsules in patients with nonvalvular atrial fibrillation.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated. Out of the 5660 enrolled subjects case report forms (CRF) were collected for 5565 subjects. It was pre-specified to combine the dose groups into one arm as the objective is to confirm appropriate use and safety profile of Prazaxa® in a real-world setting and not to compare between different dose groups.
Period: Overall Study
Arm/Group | Patients With Nonvalvular Atrial Fibrillation (NVAF)
Started (CRF collected) | 5565
Safety Set 1 | 5436
Completed | 3238
Not Completed | 2327
Not completed — Adverse Event | 480
Not completed — No actual visit | 120
Not completed — Registration rule not followed | 4
Not completed — Patients received Prazaxa treatment before | 5
Not completed — Other personal reason | 509
Not completed — To take a contraindication/careful administration drug | 8
Not completed — Lost to follow-up (changing hospital) | 373
Not completed — Lost to follow-up (unknown reason) | 146
Not completed — To conduct invasive treatment of operation | 53
Not completed — Improvement of nonvalvular atrial fibrillation | 629

BASELINE CHARACTERISTICS:
Population: Safety Set 1: This patient set included all patients who were documented to take at least one dose of Prazasa® except patients who experienced with Prazaxa® treatment for the prevention of ischemic stroke and Systemic Embolism, who did not followed registration rules, who registered outside the site contract period and/or who made no visit after the entry.
Arm/Group | Patients With Nonvalvular Atrial Fibrillation (NVAF)
Number analyzed (Participants) | 5436
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1624
  Male | 3812
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Suspected Adverse Drug Reactions (ADRs)
Description: Percentage of patients with suspected adverse drug reactions (ADRs). An adverse drug reaction is defined as a response to a medicinal product which is noxious and unintended. Response in this context means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility.
  Percentages were pre-specified to be rounded to two decimal places.
Time Frame: From baseline till the last administration + 6 days. Up to 364 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Patients With Nonvalvular Atrial Fibrillation (NVAF)
Number analyzed (Participants) | 5436
Percentage of participants | 10.69

ADVERSE EVENTS:
Time Frame: From baseline till the last administration + 6 days. Up to 364 days.
Description: Safety Set 1: all patients who took at least one dose of Prazasa® except patients who were treated with Prazaxa® for the prevention of ischemic stroke and Systemic Embolism, who did not followed registration rules, who registered outside the site contract period and/or who made no visit after entry. It was pre-specified to combine the dose groups into one arm as the objective is to confirm appropriate use and safety of Prazaxa® in a real-world setting and not comparing different dose groups.
Arm/Group | Patients With Nonvalvular Atrial Fibrillation (NVAF)
All-Cause Mortality (participants affected / at risk) | 51/5436
Serious Adverse Events (participants affected / at risk) | 416/5436
Other Adverse Events (participants affected / at risk) | 0/5436
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Nonvalvular Atrial Fibrillation (NVAF) (N=5436)
Pneumonia bacterial (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 2
Pyelonephritis acute (Infections and infestations) | 2
Bacteraemia (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Endophthalmitis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Necrotising fasciitis (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Pyelitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tuberculous pleurisy (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Arthritis infective (Infections and infestations) | 1
Infective spondylitis (Infections and infestations) | 1
Bacterial prostatitis (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Complicated appendicitis (Infections and infestations) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Angiocentric lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Basedow's disease (Endocrine disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Marasmus (Metabolism and nutrition disorders) | 1
Delirium (Psychiatric disorders) | 2
Cerebral infarction (Nervous system disorders) | 31
Embolic cerebral infarction (Nervous system disorders) | 6
Epilepsy (Nervous system disorders) | 5
Haemorrhagic cerebral infarction (Nervous system disorders) | 4
Cerebral artery embolism (Nervous system disorders) | 3
Cerebral haemorrhage (Nervous system disorders) | 3
Embolic stroke (Nervous system disorders) | 3
Cerebrovascular accident (Nervous system disorders) | 2
Dementia (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 2
Lacunar infarction (Nervous system disorders) | 2
Altered state of consciousness (Nervous system disorders) | 1
Brain stem infarction (Nervous system disorders) | 1
Cerebral atrophy (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Facial paralysis (Nervous system disorders) | 1
Myelopathy (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paralysis (Nervous system disorders) | 1
Paraparesis (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Visual field defect (Nervous system disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Carotid artery dissection (Nervous system disorders) | 1
Cerebral disorder (Nervous system disorders) | 1
Glaucoma (Eye disorders) | 2
Cataract (Eye disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Cardiac failure (Cardiac disorders) | 64
Atrial fibrillation (Cardiac disorders) | 28
Cardiac failure congestive (Cardiac disorders) | 13
Angina pectoris (Cardiac disorders) | 10
Sinus node dysfunction (Cardiac disorders) | 8
Acute myocardial infarction (Cardiac disorders) | 5
Cardiac tamponade (Cardiac disorders) | 5
Cardiac failure acute (Cardiac disorders) | 4
Atrial thrombosis (Cardiac disorders) | 4
Atrioventricular block complete (Cardiac disorders) | 3
Cardiac failure chronic (Cardiac disorders) | 3
Pericardial effusion (Cardiac disorders) | 3
Aortic valve stenosis (Cardiac disorders) | 2
Atrial flutter (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Pericardial haemorrhage (Cardiac disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 2
Aortic valve incompetence (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Bundle branch block left (Cardiac disorders) | 1
Cardiomegaly (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Sinus arrest (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia paroxysmal (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 5
Circulatory collapse (Vascular disorders) | 3
Deep vein thrombosis (Vascular disorders) | 3
Arterial occlusive disease (Vascular disorders) | 3
Embolism arterial (Vascular disorders) | 2
Haemorrhagic infarction (Vascular disorders) | 2
Aortic aneurysm (Vascular disorders) | 1
Aortic aneurysm rupture (Vascular disorders) | 1
Aortic dissection (Vascular disorders) | 1
Arteriovenous fistula (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
Arterial stenosis (Vascular disorders) | 1
Atheroembolism (Vascular disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6
Melaena (Gastrointestinal disorders) | 4
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 3
Mechanical ileus (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Pancreatitis acute (Gastrointestinal disorders) | 2
Rectal ulcer (Gastrointestinal disorders) | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Large intestine polyp (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastric dilatation (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastric hypomotility (Gastrointestinal disorders) | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Large intestinal stenosis (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 3
Acute hepatic failure (Hepatobiliary disorders) | 2
Cholangitis (Hepatobiliary disorders) | 2
Cholangitis acute (Hepatobiliary disorders) | 2
Drug-induced liver injury (Hepatobiliary disorders) | 2
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hepatitis fulminant (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Primary biliary cholangitis (Hepatobiliary disorders) | 1
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 6
Renal impairment (Renal and urinary disorders) | 3
Renal failure (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Calculus urinary (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal infarct (Renal and urinary disorders) | 1
Postrenal failure (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2
Prostatic haemorrhage (Reproductive system and breast disorders) | 1
Death (General disorders) | 6
Chest discomfort (General disorders) | 2
Sudden death (General disorders) | 2
Chest pain (General disorders) | 1
Generalised oedema (General disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Oedema due to cardiac disease (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Heart rate decreased (Investigations) | 1
Weight increased (Investigations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 5
Fall (Injury, poisoning and procedural complications) | 4
Pelvic fracture (Injury, poisoning and procedural complications) | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1
Finger amputation (Surgical and medical procedures) | 1
Mitral valve replacement (Surgical and medical procedures) | 1
Valvuloplasty cardiac (Surgical and medical procedures) | 1
Cardiac ablation (Surgical and medical procedures) | 1
Cardiac operation (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT03175198/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT03175198/SAP_001.pdf